CLINICAL TRIAL: NCT06607302
Title: Ivosidenib in Locally Advanced or Metastatic Cholangiocarcinoma With IDH1 R132 Mutation After at Least One Prior Systemic Treatment - a Prospective, Multicenter, Observational Study in Germany
Brief Title: Ivosidenib in Locally Advanced or Metastatic Cholangiocarcinoma With IDH1 R132 Mutation After at Least One Prior Systemic Treatment - an Observational Study
Acronym: IDHIRA
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Servier Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: iOM-040498
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Storage location of tumor samples collected during clinical routine will be documented within a virtual biobank
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cholangiocarcinoma is a rare and aggressive tumor of the bile duct associated with a poor prognosis and very limited treatment options. The IDH1 inhibitor ivosidenib provides a new, targeted treatment option for this disease. Ivosidenib was approved by European Medicines Agency (EMA) in May 2023 as monotherapy in adult patients with locally advanced or metastatic cholangiocarcinoma with an IDH1 R132 mutation who were previously treated by at least one prior line of systemic therapy.

The prospective, multicenter, observational study IDHIRA will collect first real-world data on ivosidenib treatment in a broad patient population in Germany. Ivosidenib will be administered according to the current SmPC. Thus, IDHIRA will generate real-world evidence on effectiveness, quality of life (QoL) and safety of ivosidenib.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Histologically confirmed locally advanced or metastatic CCC with a documented IDH1 R132 mutation diagnosed by an appropriate diagnostic test
* Patients must have at least one prior systemic therapy
* Decision for treatment with ivosidenib according to current SmPC.
* Signed written informed consent before or within 6 weeks of first ivosidenib dose (inclusion of patients up to 6 weeks after first ivosidenib intake is allowed for patients not participating in the PRO module)
* For patients participating in the PRO module (optional):

  * Dated signature of informed consent form before start of study treatment.
  * Willingness and capability to participate in PRO assessment in German language.
* Other criteria according to current SmPC.

Exclusion Criteria:

* Participation in an interventional clinical trial within 30 days prior to enrolment or concurrent participation in an interventional clinical trial except for the follow-up period.
* Other contraindications according to current SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IDH1 R132-mutated locally advanced or metastatic CCC who have received at least one prior line of systemic therapy and who have already been scheduled by their treating physician to receive ivosidenib prior to enrolment in IDHIRA are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | max. 38 months (FPI - LPLV)
  PFS is defined as the time interval measured from the day of first ivosidenib administration to first progression or death, whichever comes first. Patients without tumor progression or death at the time of analysis will be censored at their date of last contact.

SECONDARY OUTCOMES:
Overall survival (OS) | max. 38 months (FPI - LPLV)
  OS is defined as the time interval measured from the day of first ivosidenib administration to time of death from any cause. Time to last contact will be used if a patient has no documented date of death and OS for the patient will be considered censored.
Timt to treatment failure (TTF) | max. 38 months (FPI - LPLV)
  TTF is defined as the time interval measured from the day of first ivosidenib until discontinuation of treatment for any reason including progression, toxicity, start of a new antineoplastic therapy, or death, whichever occurs first. Patients dropping out without knowledge of a potential ending of therapy (e.g., lost to follow up) will be censored with the last date of contact.
Overall response rate (ORR) | max. 38 months (FPI - LPLV)
  ORR is defined as the proportion of patients achieving a complete or partial response as best response. Patients without response measurement are considered non-responders.
Disease control rate (DCR) | max. 38 months (FPI - LPLV)
  DCR is defined as the proportion of patients achieving complete response, partial response, or stable disease as best response. Patients without response measurement are considered non-responders.
(Serious) adverse events ((S)AE)) | max. 38 months (FPI - LPLV)
  The case- and patient-based incidence of (S)AEs will be provided.
(Serious) adverse drug reactions ((S)ADR) related to ivosidenib | max. 38 months (FPI - LPLV)
  The case- and patient-based incidence of (S)ADRs will be provided.
Adverse events of special interest (AESI) | max. 38 months (FPI - LPLV)
  The case- and patient-based incidence of AESIs will be provided.
Global health-related quality of life during course of treatment | max. 38 months (FPI - LPLV)
  The change from baseline (i.e., difference) in the scales of the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer quality of life questionnaire C30) will be displayed for each point in time, using boxplots.
  The scales of the EORTC QLQ-C30 range in score from 0 to 100. A high scale score represents a higher response level.
Cholangiocarcinoma-related quality of life during course of treatment | max. 38 months (FPI - LPLV)
  The change from baseline (i.e., difference) in the scales of the EORTC QLQ-BIL21 (European Organisation for Research and Treatment of Cancer quality of life questionnaire BIL21) will be displayed for each point in time, using boxplots.
  The scales of the EORTC QLQ-BIL21 range in score from 0 to 100. A high scale score represents a higher response level.
Assessing parameters of physician treatment decision making | max. 30 months (recruitment period)
  Frequencies of distinct impact ratings for parameters affecting ivosidenib therapy choice will be visualized using stacked bar charts.
Assessing parameters of physician treatment satisfaction | max. 32 months (recruitment period plus 8 weeks)
  Frequencies of distinct satisfaction levels with ivosidenib treatment effectiveness and AE management will be visualized using stacked bar charts.
Cumulative ivosidenib dose | max. 38 months (FPI - LPLV)
  Summary tables containing descriptive statistics (n, mean, standard deviation, median, 25th and 75th percentiles, minimum, and maximum) will be provided.
Absolute dose intensity of ivosidenib | max. 38 months (FPI - LPLV)
  Summary tables containing descriptive statistics (n, mean, standard deviation, median, 25th and 75th percentiles, minimum, and maximum) will be provided.
Relative dose intensity of ivosidenib | max. 38 months (FPI - LPLV)
  Summary tables containing descriptive statistics (n, mean, standard deviation, median, 25th and 75th percentiles, minimum, and maximum) will be provided.
Frequency of dose modifications | max. 38 months (FPI - LPLV)
  Frequency of dose modifications will be presented.
Type of dose modifications | max. 38 months (FPI - LPLV)
  Type of dose modifications (i.e., dose reductions, dose escalations, and interruptions) will be presented.
Reasons for dose modifications | max. 38 months (FPI - LPLV)
  Reasons for dose modifications will be presented.
Duration of treatment with ivosidenib | max. 38 months (FPI - LPLV)
  Duration of treatment with ivosidenib
Reasons for end of treatment (EOT) | max. 38 months (FPI - LPLV)
  Reasons for end of treatment will be displayed
Type of last previous therapy | max. 38 months (FPI - LPLV)
  Type of substances given in the last previous therapy will be displayed.
Frequency of last previous therapy | max. 38 months (FPI - LPLV)
  Frequency of different substances given in the last previous therapy will be displayed.
Duration of last previous therapy line | max. 38 months (FPI - LPLV)
  Duration of last previous therapy line will be displayed.
Concomitant medications | max. 38 months (FPI - LPLV)
  Frequency of concomitant medications in total will be displayed.
Concomitant medications known to induce QT prolongation | max. 38 months (FPI - LPLV)
  Frequency of concomitant medications known to induce QT prolongation (e.g., antiarrhythmic medicines, fluoroquinolones, triazole anti-fungals, 5-HT3 receptor antagonists) will be displayed.
Subsequent antineoplastic therapies | max. 38 months (FPI - LPLV)
  Frequency and type of subsequent antineoplastic therapies by line of therapy will be displayed.

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (7):
  - Hämatologisch-Onkologische Schwerpunktpraxis in Bad Liebenwerda, Bad Liebenwerda
  - Caritas Krankenhaus Bad Mergentheim, Bad Mergentheim
  - Onkologisches Versorgungszentrum Berlin MVZ, Berlin
  - Onkologie Hannover, Hanover
  - Onkologie Hof, Hof
  - Medizinisches Versorgungszentrum Mönchengladbach, Mönchengladbach
  - ze:roPRAXEN MVZ für Innere Medizin, Weinheim

REFERENCES:
- [Derived] Michl M, Hagemeyer N, Looss M, Grebhardt S, Ringwald K, Potthoff K. IDHIRA: a prospective, observational study on ivosidenib in patients with IDH1 R132-mutated advanced cholangiocarcinoma. Future Oncol. 2025 Apr;21(9):1057-1064. doi: 10.1080/14796694.2025.2470609. Epub 2025 Mar 3. PMID 40028796